CLINICAL TRIAL: NCT03449056
Title: High-flow Nasal Cannula Nebulization of Beta 2 Adrenergic Agonist During Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: OPTINEB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPTINEB
Record Dates: First submitted 2018-01-12; First posted 2018-02-28 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; High-flow Nasal Cannula
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TREATMENT (Experimental): salbutamol nebulization
  Interventions: Drug: salbutamol

INTERVENTIONS:
Drug: salbutamol — T2 - T1+1h30: High-nasal flow and salbutamol nebulization

SUMMARY:
High-flow nasal cannula is an oxygenation technique increasingly used for patients admitted for acute respiratory failure. Literature essentially concerns "de novo" acute hypoxemic failure and the interest of high-flow during take care of chronic obstructive pulmonary disease patients is few studied. Physiological studies reported potential benefits of high-flow nasal cannula oxygenation in chronic obstructive pulmonary disease patients including dead space clearance and decrease of respiratory, which lead to decrease work of breathing. As inhaled bronchodilators are part of treatment of chronic obstructive pulmonary disease exacerbation, nebulization could be also provided through high-flow nasal cannula oxygen therapy. The aim of our study is to determine whether a beta-2 agonist nebulization administered through High-flow nasal cannula is efficient to improve spirometry of patients for admitted hronic obstructive pulmonary disease exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Arterial pH over 7.25,
* Respiratory rate under 35 breaths/mn
* Glasgow Coma Scale equal to 15,
* indication of beta-2 agonist nebulization less than 8 per day (time between two nebulization more than 3 hours),
* NIV sessions spaced more than 6 hours.

Exclusion Criteria:

* Urgent endotracheal intubation;
* Contraindication to beta 2 adrenergic agonist;
* Another organ failure (hemodynamic and neurological instability);
* Cardioselective beta-blocker during treatment of copd exacerbation;

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
compare lung functions | baseline-1h30
  Evolution of Forced Expiratory Volume 1s

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No